CLINICAL TRIAL: NCT07156695
Title: Deep Marginal Elevation and Its Impact on Periodontal Microenvironment: Microbiological, Clinical, and Radiographic Study
Brief Title: Deep Marginal Elevation and the Periodontal Microenvironment ( DME-PM )
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Omar Elboraey Elbal, Assistant Professor of Oral Medicine, Periodontology, Oral Diagnosis and Oral Radiology Department, Faculty of Dentistry, Tanta, University, Tanta, Egypt., Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #R-RD-2-25-3190
Record Dates: First submitted 2025-08-25; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Deep Marginal Elevation; Periodontal Microenvironment; Microbiological Study; Clinical Study; Radiographic Study

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deep Marginal Elevation (DME) (Experimental): Participants with Class II dental caries will receive Deep Marginal Elevation (DME) using resin-modified glass ionomer cement (RMGIC) followed by adhesive and nano filled composite restoration.
  Interventions: Procedure: Deep Marginal Elevation (DME)

INTERVENTIONS:
Procedure: Deep Marginal Elevation (DME) — Deep Marginal Elevation (DME) is performed by elevating the deep margin of Class II cavities using resin-modified glass ionomer cement (RMGIC), followed by adhesive bonding and placement of a nanofilled composite resin restoration. This procedure improves accessibility of the restorative margin, enhances marginal sealing, and facilitates plaque control.

SUMMARY:
This study aims to evaluate the impact of the dental restorative procedure known as Deep Marginal Elevation (DME) on periodontal health, including gingival and bone status, in patients with deep dental caries. Gingival fluid samples will be collected, and radiographic assessments will be performed to monitor changes in inflammation and bone levels. The findings are expected to provide insights into how DME influences gingival and bone health.

DETAILED DESCRIPTION:
Deep Marginal Elevation (DME) represents a significant advancement in restorative dentistry, providing a promising solution for the management of deep caries lesions, particularly in Class II cavities. The technique involves elevating the deep margin of the cavity to a more accessible level, thereby facilitating placement of a durable restoration while preserving pulp vitality.

Despite increasing adoption in clinical practice, the impact of DME on the periodontal microenvironment-specifically its influence on inflammatory and microbiological markers-remains insufficiently explored.

Inflammatory markers such as Interleukin-1β (IL-1β), Tumor Necrosis Factor-alpha (TNF-α), Matrix Metalloproteinase-8 (MMP-8), Prostaglandin E2 (PGE2), and C-Reactive Protein (CRP) play pivotal roles in the pathogenesis of periodontal disease. Monitoring these biomarkers in gingival crevicular fluid (GCF) provides valuable insights into the inflammatory status of periodontal tissues.

In addition to inflammatory markers, bone level and bone density serve as critical indicators of periodontal health, with alterations often reflecting disease progression. Bitewing radiographs offer a reliable method for assessing these parameters.

This investigation is designed as a longitudinal clinical study to evaluate the effects of DME on GCF microbiological and inflammatory markers, as well as bone level, crestal bone loss, and bone density.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-60 years.
* Diagnosed with Class II dental caries requiring restoration.
* Presence of a healthy contralateral tooth (control side).
* Willingness to participate and comply with follow-up visits.

Exclusion Criteria:

* Systemic diseases (e.g., diabetes, autoimmune disorders).
* Periodontal disease or active infection.
* Use of anti-inflammatory medications within the last month.
* Pregnancy or lactation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Gingival Crevicular Fluid (GCF) Microbiological Markers | 1 month post-intervention.
  Assessment of microbial load in GCF samples to evaluate the microbiological impact of Deep Marginal Elevation will be recorded at the baseline, immediately post-intervention, and 1 month post-intervention.

SECONDARY OUTCOMES:
Changes in Gingival Crevicular Fluid (GCF) Inflammatory Markers | 1 month post-intervention.
  Measurement of cytokines (IL-1β, TNF-α, MMP-8, PGE2, CRP) in GCF samples to assess the inflammatory periodontal response to Deep Marginal Elevation will be recorded at the baseline, immediately post-intervention, and 1 month post-intervention.
Changes in Bone Level | 1 month post-intervention.
  Evaluation of the distance from the cementoenamel junction (CEJ) to the alveolar crest on standardized bitewing radiographs will be recorded at the baseline, immediately post-intervention, and 1 month post-intervention.
Changes in Crestal Bone Loss | 1 month post-intervention.
  Quantification of crestal bone height reduction associated with the intervention using standardized bitewing radiographs will be recorded at the baseline, immediately post-intervention, and 1 month post-intervention.
Changes in Bone Density | 1 month post-intervention.
  Grayscale analysis of alveolar bone density from standardized bitewing radiographs will be recorded at the baseline, immediately post-intervention, and 1 month post-intervention.
Changes in Gingival Index (GI) | 1 month post-intervention.
  Evaluation of gingival inflammation severity will be performed using the Gingival Index (GI) . This index scores gingival tissues based on color, consistency, and bleeding on probing.
  Scale Details:
  Range: 0 to 3
  0 = Normal gingiva (no inflammation)
  1. = Mild inflammation (slight color change, slight edema, no bleeding on probing)
  2. = Moderate inflammation (redness, edema, glazing, bleeding on probing)
  3. = Severe inflammation (marked redness and edema, ulceration, spontaneous bleeding) Direction of Scoring: Higher scores indicate worse gingival inflammation.
Changes in Bleeding Index (BI) | 1 month post-intervention.
  Assessment of gingival bleeding tendency on probing will be performed using the Bleeding Index (BI). This index evaluates the presence or absence of bleeding as an indicator of gingival inflammation.
  Scale Details:
  Range: 0 to 1
  0 = No bleeding on probing
  1 = Bleeding on probing present Direction of Scoring: Higher scores indicate worse gingival inflammation.
Changes in Clinical Attachment Loss (CAL) | 1 month post-intervention.
  Periodontal attachment level will be assessed using a manual periodontal probe to measure the distance (in millimeters) from the cementoenamel junction (CEJ) to the base of the gingival sulcus/pocket. Measurements will be taken at baseline, immediately post-intervention, and at 1-month follow-up to evaluate periodontal tissue stability after Deep Marginal Elevation (DME).
  Scale/Units:
  Measurement tool: Periodontal probe (UNC-15)
  Range: 0 mm to 15 mm (probe scale)
  Interpretation:
  Lower clinical Attachment Loss (CAL) values = better periodontal attachment and stability
  Higher CAL values = greater tissue destruction and worse periodontal health
  Direction of Scoring: Higher CAL values indicate worse periodontal outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author